CLINICAL TRIAL: NCT05575440
Title: Evaluation of F-18 Tetrafluoroborate (18F-TFB) PET/CT in Patients With Differentiated Thyroid Cancer
Brief Title: Evaluation of 18F-TFB PET/CT Scan in Patients With Differentiated Thyroid Cancer
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 20-010573; NCI-2022-03071 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Differentiated Thyroid Gland Carcinoma; Thyroid Gland Follicular Carcinoma; Thyroid Gland Papillary Carcinoma
MeSH Terms: conditions — Adenocarcinoma, Follicular; Thyroid Cancer, Papillary | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (18F-TFB PET/CT): Patients receive fluorine F18 tetrafluoroborate IV and undergo PET/CT scan on study.
  Interventions: Procedure: Computed Tomography; Radiation: Fluorine F 18 Tetrafluoroborate; Procedure: Positron Emission Tomography; Other: Survey Administration

INTERVENTIONS:
Procedure: Computed Tomography — Undergo a PET/CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Radiation: Fluorine F 18 Tetrafluoroborate — Given IV
  Other Names: 18F-Tetrafluoroborate; 18F-TFB
Procedure: Positron Emission Tomography — Undergo a PET/CT scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Other: Survey Administration — Ancillary studies

SUMMARY:
This phase II study evaluates F-18 tetrafluoroborate (18F-TFB) PET/CT scan in patients with differentiated thyroid cancer. Diagnostic imaging is necessary for planning treatment, monitoring therapy response, and identifying sites of recurrent or metastatic disease in differentiated thyroid cancer. 18F-TFB PET/CT may accurately detect recurrent and metastatic thyroid cancer lesions, with the potential to provide information for patient management that is better than the current standard of care imaging practices.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate fluorine F 18 tetrafluoroborate (18F-TFB) positron emission tomography (PET)/computed tomography (CT) imaging in patients with intermediate or high risk differentiated thyroid cancer (DTC) and compare to the current clinical standard.

II. Assess the impact of 18F-TFB PET/CT on clinical management.

OUTLINE:

Patients receive fluorine F 18 tetrafluoroborate intravenously (IV) and undergo PET/CT scan on study.

ELIGIBILITY:
Inclusion Criteria:

* Subject has biopsy-proven papillary or follicular thyroid cancer
* Subject is clinically indicated for 123I-SPECT/CT total body iodine (TBI) scan
* Subject agrees to undergo 18F-TFB PET/CT scan following TBI scan
* Karnofsky performance status of >= 50 (or Eastern Cooperative Oncology Group [ECOG]/World Health Organization [WHO] equivalent)
* Subject is able to be scanned - able to lie still on SPECT/CT and PET/CT scanner table for up to 65 minutes (min)
* Age 18 or older
* Ability to understand a written informed consent document, and the willingness to sign it
* Subject is not pregnant

Exclusion Criteria:

* Contrast-enhanced CT within 4 last weeks
* Amiodarone within last 4 months
* Ingested iodine, kelp tablets, Lugols iodine, or potassium iodide (SSKI) within 2 weeks
* Unable to lie flat, still or tolerate a PET scan
* Applied betadine, iodoform, or quick tanning products to skin within last two weeks
* If using medication withdrawal for stimulation, then exclude if thyroid stimulating hormone (TSH) level < 25
* Taken anti-thyroid medication within 1 week
* Subject is breastfeeding
* Positive pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects have biopsy-proven papillary or follicular thyroid cancer and is clinically indicated for 123I-single-photon emission computerized tomography (I-SPECT)/CT total body iodine (TBI) scan
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Descriptive summaries of detected lesions | Up to 2 years
  Descriptive summaries of detected lesions (presence/absence) will include counts and proportions at the patient and lesion level. Overall concordance of these measures across modalities will be estimated using Cohen's kappa with 95% confidence intervals generated by clustered bootstrapping. Per-lesion analysis of detection rates by modality will be performed using cluster-adjusted McNemar's test, accounting for the paired nature of the data (i.e., two scans) and potential within-sample correlation for patients with multiple lesions.
Conspicuities and diagnostic confidence scores for a given lesion | Up to 2 years
  Conspicuities and diagnostic confidence scores for a given lesion will be averaged across readers. Descriptive summaries of these scores will include medians and interquartile ranges. Concordance of these measures across modality will be evaluated using Lin's concordance correlation coefficient with 95% confidence intervals generated by clustered bootstrapping. Differences in conspicuities and diagnostic confidence scores will be tested using cluster-adjusted Wilcoxon signed-rank tests.

SECONDARY OUTCOMES:
True positive and negative lesions | Up to 2 years
  Given true positive and negative lesions determined by histopathology and/or imaging, clinical and laboratory follow-up, we will estimate sensitivity, specificity, net present value, and positive predictive value on a per-lesion and patient basis for 18F TFB PET/CT and 123I single-photon emission computerized tomography/CT along with the corresponding two-sided 95% confidence intervals. The confidence intervals will be constructed using clustered bootstrapping.
Impact of PET on clinical management in differentiated thyroid cancer (DTC) patients | Up to 2 years
  The impact of PET on clinical management in DTC patients will be evaluated using descriptive statistics. Evidence of discordance among the modalities will be assessed using a McNemar- Bowker test of symmetry.
Inter-reader reproducibility | Up to 2 years
  Inter-reader reproducibility will be assessed for positivity at the patient level and region level (nominal) as well as standardized uptake values (SUVs) for positive lesions (quantitative). Reproducibility will be reported using the Fleiss' Kappa test for multiple readers for positivity and Pearson intra-class correlation for SUVs.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M. Broski, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials